CLINICAL TRIAL: NCT02217748
Title: Understanding Name Generator Order Effects When Eliciting Social Networks in Rural Uganda: A Randomized Controlled Trial
Brief Title: Name Generator Order Effects in Social Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MH096620-S2
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Social Interaction
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Survey questionnaire version 1 (Experimental): Name generator order: leisure, money, support
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 2 (Experimental): Name generator order: leisure, support, money
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 3 (Experimental): Name generator order: money, leisure, support
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 4 (Experimental): Name generator order: money, support, leisure
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 5 (Experimental): Name generator order: support, leisure, money
  Interventions: Other: Survey questionnaire
- Survey questionnaire version 6 (Experimental): Name generator order: support, money, leisure
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire
  Other Names: Each of the survey questionnaires administers the name generators in a different order

SUMMARY:
The objective of our study was to determine the extent to which the order of specific items in a multiple name generator survey affects how social networks are measured.

DETAILED DESCRIPTION:
Interpersonal relationships are one feature of the social environment that have been shown to have important influences on health and health behaviors (Berkman et al., 2000; Berkman & Syme, 1979) and mental health (Tsai et al., 2014). While the majority of these studies have been conducted in resource-rich settings, studies conducted in resource-limited settings have similarly demonstrated associations between social networks and health (Perkins, Subramanian, & Christakis, 2014). In this literature, the tie between two persons is the important unit of measurement. Classically, the social tie is typically elicited using a "name generator" survey that inquires about ties based on the affective content of the relationship (Laumann, 1966; Wellman, 1979) or normative bonds such as kinship ties (Kleiner & Parker, 1976).

Another popular approach to eliciting social ties has employed multiple name generators inquiring about specific types of interactions, such as discussions about important matters or exchanges of money (Burt, 1984; Marsden, 1987; McCallister & Fischer, 1978). These types of name generators have strong face validity, are less likely to be subjectively interpreted in different ways by different respondents, and are therefore likely to be more reliable. These are accompanied by a heavy respondent burden, however, and single-item name generators may perform comparably to multiple name generators only under limited circumstances (Marin & Hampton, 2007). It remains unclear, however, whether the order of name generators may affect study participant responses. While no studies have examined this empirically, there is a broad literature on public opinion polling suggesting that alternative specifications of question ordering can have important effects on respondents' answers (McFarland, 1981).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Emancipated minors aged 16-18 years
* Considers Nyakabare Parish their primary place of residence
* Capable of providing informed consent

Exclusion Criteria:

* Minors younger than 18 years, with the exception of emancipated minors
* Does not consider Nyakabare Parish their primary place of residence
* Unable to communicate with research staff, e.g., due to deafness, mutism, or aphasia
* Persons with psychosis, neurological damage, acute intoxication, or an intelligence quotient less than 70, as determined in the field by non-clinical research staff in consultation with a supervisor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1557 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of social ties elicited by a specific name generator | Baseline
Number of social ties elicited by the composite name generator | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital; Bernard Kakuhikire, MBA, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda